CLINICAL TRIAL: NCT02115503
Title: A Prospective, Global, Multi-center, Treatment Registry Study of Intravenous Immunoglobulin Maintenance Therapy in Alloantibody Positive Renal Allograft Recipients
Acronym: DSA
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Databean (Industry)
Collaborators: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: DSA 3242014
Record Dates: First submitted 2014-04-04; First posted 2014-04-16 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Renal Transplant Recipients With Anti-HLA Antibodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort 1: Cohort 1 will consist of those having primarily Class I antibody development post-transplant
- Cohort 2: Cohort 2 will include those having primarily Class II antibody development post-transplant
- Cohort 3: Cohort 3 will consist of the remaining subjects that have a mix of Class I and II antibodies.

SUMMARY:
The purpose of this treatment registry study is to determine if monthly infusions of Intravenous Immunoglobulin (IVIg) for 6 months will neutralize donor specific antibodies that are thought to be responsible for chronic rejection episodes in renal transplant subjects. 162 renal transplant subjects will receive IVIg 5% at 2gm/kg/month for 6 months and be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Able to provide voluntary written informed consent
* Renal transplant recipient at least 1 month post-transplant
* On stable doses of maintenance immunosuppression for at least 14 days prior to study entry and remains on stable maintenance doses for the duration of the study
* Presence of DSA greater than or equal to 1000 mean fluorescence intensity (MFI) single antigen bead assay via Luminex (normalized 2,000 - 15,000 MFI, inclusive) measured within 6 months prior to consent
* Female subjects must be post-menopausal for at least 1 year, or surgically sterilized, or must agree to use two effective methods of birth control from the time of consent through 30 days after the last dose of IVIg.
* Male subjects must be surgically sterilized, or must agree to use two effective methods of birth control from the time of consent through 30 days after the last dose of IVIg
* Subject is compliant and intends to be available for follow-up study period of 3 years

Exclusion Criteria:

* Multi-organ transplant
* History of anaphylactic or severe systemic reactions to human immunoglobulin
* IgA deficient subjects with antibodies against IgA and a history of hypersensitivity
* Serum creatinine > 3.0 mg/dL within 90 days prior to consent
* Recipients of ABO incompatible kidney transplants
* Acute rejection within 180 days (6 months) prior to consent defined as:

  1. Biopsy proven acute Cellular Rejection [Banff grade I (including IA and IB), grade II (including IIA and IIB) or grade III]; or
  2. an antibody-mediated rejection with C4d positivity, or
  3. chronic rejection with C4d positivity (C4d positivity is defined as staining diffuse in peritubular capillary area. Isolated C4d glomerular staining or C4d staining of < 50% of the peritubular capillaries will not be exclusion criteria). Borderline cellular rejection will not be excluded (Banff 2005), or
  4. Clinical signs and symptoms of acute rejection including elevated creatinine, fever over 100 degrees, pain or tenderness around the transplanted kidney, fluid retention of the hands, legs, feet, ankles or eyelids, sudden weight gain (2-4 pounds in a day, or 5 pounds or more in a week), decrease in urine output with the same amount of fluid intake, or dark yellow or orange urine output, flu-like symptoms, such as chills, aches, tiredness, dizziness, nausea, loss of appetite, weakness, fatigue, vomiting or general sense of not feeling well (Note: NOT all signs and symptoms need to be present to document acute rejection)
* Evidence of proteinuria (> 3 grams) within 90 days (3 months) prior to consent
* Active CMV+ or EBV+ viremia that requires, or will require, anti-viral therapy
* History of HCV, HIV and/or HBsAg positivity
* History of post-transplant lymphoproliferative disease.
* Active BK/polyomavirus nephropathy, or BK/polyomavirus nephritis that requires, or will require, anti-viral therapy (not prophylactic)
* Recipients of a kidney from a donor who tests positive for HIV, HBsAg or anti-HCV.
* History of malignancy within the past 5 years that is not considered to be cured, with the exception of complete resection of localized basal cell carcinoma of the skin (excised ≥ 1 years prior to enrollment).
* Subjects who are receiving everolimus, sirolimus or azathioprine as immunosuppressive agents and who are unwilling, or unable, to change to mycophenolate mofetil or mycophenolic acid within 14 days prior to consent
* White blood cell count of <1,000/mm3 within 90 days prior to consent
* Platelet count <60,000/mm3 within 90 days prior to consent
* Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3 times upper limit of normal [ULN]) within 90 days prior to consent
* Total bilirubin > 1.5 times ULN within 90 days prior to consent
* Post-transplant history of cardiovascular disease within 180 days (6 months) prior to consent defined as:

  1. Electrocardiographic evidence of MI,
  2. Electrocardiographic evidence of acute ischemia,
  3. Electrocardiographic evidence of severe conduction system abnormalities OR
  4. New York Heart Association (NYHA) Class II - IV heart failure (Subjects with other cardiac abnormalities may be included if documented by the investigator as not clinically significant)
* Pregnant or nursing (lactating) women
* Enrolled in any other treatment study within 30 days of consent
* Serious medical illness (other than renal disease), or psychiatric illness likely to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-07; Primary Completion 2019-08 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Difference in mean change from screening to 36 months in graft survival and glomerular filtration rates (GFR) | 3 years
  Success is defined as:
  Allograft survival as compared to the performance goal (PG) at 36 months. For the purposes of this study, a graft will be presumed to be lost is when a subject is started on dialysis and is not able to subsequently be removed from dialysis; or a subject's serum creatinine reaches 4.0 mg/dL, is sustained for >48hours and is not thought to be due to other causes; or the subject is re-transplanted; or the subject dies. AND:
  A change in extended GFR, defined as <15% decrease in mean GFR from baseline to 36 months

SECONDARY OUTCOMES:
Allograft Survival | 3 years

OTHER OUTCOMES:
Allograft survival in subjects with preformed DSA defined as an MFI > 500 at the time of transplantation | 3 years
Allograft survival in subjects who are recipients of >1 renal transplant | 3 years
A difference in mean change of extended GFR ml/min/1.73 m2 (eGFR - MDRD) | 3 years
Incidence of proteinuria (urine protein:creatinine > 1.5) at 1, 2 and 3 years | 3 years
Change in proteinuria from screening to 1, 2, and 3 years | 3 years
Change in serum creatinine from screening to 1, 2, and 3 years | 3 years
Proportion of subjects that achieve a complete response defined as a return of DSAmax antibody MFI to less than 2000 at 9 months | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: A. O. Gaber, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (8):
- United States (8):
  - St Vincent's Transplant Research Institute, Los Angeles, California
  - University of California Davis Health Systems, Sacramento, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cornell Medical Center, New York, New York
  - Baylor Research Institute, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas